CLINICAL TRIAL: NCT06012786
Title: Myofascial Pain Syndrome in Patients With Breast Cancer-related Lymphedema
Status: Completed | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 23/338
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Myofascial Pain Syndrome; Breast Cancer; Breast Cancer Female; Lymphedema; Lymphedema of Upper Limb; Pain
Keywords: breast cancer; myofascial pain syndrome; lymphedema
MeSH Terms: conditions — Myofascial Pain Syndromes; Breast Neoplasms; Lymphedema; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (Patients with Stage 0 lymphedema): It is known that pathophysiological changes develop even if there is no visible lymphedema in patients undergoing surgery and/or radiotherapy for breast cancer. There is a lifetime risk of developing lymphedema, so these patients are considered as Stage 0 (latent). The patients with less than 3 cm difference between the circumference measurements of upper extremities will be included in the 1st group.( Stage 0) (n=55)
  Interventions: Diagnostic Test: Diagnostic Criteria of Myofascial Pain Syndrome; Diagnostic Test: The Physical Examination of Trigger Points and Pain-Pressure Threshold Measurement With an Algometer; Diagnostic Test: Hand Grip Test; Diagnostic Test: VAS; Diagnostic Test: Quick DASH; Diagnostic Test: Lymqol-Arm; Diagnostic Test: Range of Motion of Shoulde Joint
- Group 2 (Patients with Stage 1,2 or 3 lymphedema): Patients who have more than 3 cm difference between the circumference measurements of upper extremities and those with Stage 1,2 or 3 lymphedema will be included in the second group (n=55)
  Interventions: Diagnostic Test: Diagnostic Criteria of Myofascial Pain Syndrome; Diagnostic Test: The Physical Examination of Trigger Points and Pain-Pressure Threshold Measurement With an Algometer; Diagnostic Test: Hand Grip Test; Diagnostic Test: VAS; Diagnostic Test: Quick DASH; Diagnostic Test: Lymqol-Arm; Diagnostic Test: Range of Motion of Shoulde Joint

INTERVENTIONS:
Diagnostic Test: Diagnostic Criteria of Myofascial Pain Syndrome — Major criteria:
  1. The patient's complaint of regional pain
  2. Referred pain and sensory change in the specific area of the muscle by palpation of the trigger point
  3. Presence of palpable taut band
  4. Presence of palpable and tender points along the length of the taut band
  5. Restriction of ROM in the area of the affected muscle
  Minor criteria:
  1. Pain/sensory change with pressure palpation of the trigger point
  2. Local twitch response with palpation/injection of the trigger point in the taut band
  3. Reduction of pain by inactivation (injection or stretching of the muscle) of the trigger point 5 major and at least 1 minor criteria are required for clinical diagnosis
Diagnostic Test: The Physical Examination of Trigger Points and Pain-Pressure Threshold Measurement With an Algometer — Trigger points in trapezius, infraspinatus, latissimus dorsi, pectoralis major, serratus anterior muscles will be detected bilaterally by physical examination. Algometer (Wagner Force Dial FDK 20) will be used for pain pressure threshold measurement of detected trigger points. Then, the distribution of the trigger points, their frequency and threshold values according to the algometer will be compared between the individual affected-insured extremities and between the groups.
Diagnostic Test: Hand Grip Test — The purpose of this test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer (Jamar) will be used for the test. While the patient is sitting in the chair, the elbows will be close to the body and at 90 degree flexion, the wrist will be in a neutral position. The patient will be asked to grasp the dynamometer and squeeze it as hard as she can, and the average of 3 measurements made with an interval of 5 minutes. The test will be repeated for both upper extremities separately.
Diagnostic Test: VAS — Shoulder pain, feeling of tension and heaviness on the affected arm will be evaluated separately by numerical scale.
Diagnostic Test: Quick DASH — The quick DASH questionnaire which has proven reliable and valid in breast cancer and lymphedema patients in Turkish population, will be used to evaluate the quality of life related to upper extremity function.
Diagnostic Test: Lymqol-Arm — Lymphedema Quality of Life Scale-Arm Turkish form will be used. The lymphedema-specific quality of life scale was developed specifically for the upper extremity and its reliability and validity were proven in Turkish population.
Diagnostic Test: Range of Motion of Shoulde Joint — Goniometric measurements will be made for both upper extremities, and the average of 3 consecutive measurements will be taken.

SUMMARY:
The goal of this observational study is to determine the relationship between Lymphedema and Myofascial Pain Syndrome in Breast Cancer Patients.

The main questions it aims to answer:

* Is there a relationship between the stage of lymphedema and the frequency of accompanying myofascial pain syndrome in the breast cancer patients?
* Does the existence of lymphedema in breast cancer patients affect the distribution and the pain threshold values of trigger points seen in Myofascial Pain Syndrome?
* What is the impact of Myofascial pain syndrome seen in breast cancer associted lymhedema patients on upper extremity function and quality of life?

DETAILED DESCRIPTION:
Mastectomy, breast conserving surgery, axillary lymph node dissection, sentinel lymph node biopsy and radiotherapy treatments have significant results in skin, muscle and fascia tissues in the upper extremity.

Upper extremity function is defined by the International Consortium for Measures of Health Outcomes (ICHOM) as one of the most important health measures in breast cancer patients. Long-term upper extremity dysfunction has serious effects on patients' quality of life.

Lymphedema, severe pain, decrease in shoulder joint range of motion, myofascial pain syndrome, myofascial adhesions are the leading causes affecting upper extremity function in patients with breast cancer.

Myofascial pain syndrome (MPS) is commonly seen in patients with musculoskeletal problems and originates from muscle and surrounding tissues. It is characterized by localized or referred pain in a limited area and trigger points in the affected muscles. The incidence of myofascial pain syndrome secondary to breast cancer surgery is unknown. There is not yet a study in the literature that reveals the relationship between the stage of lymphedema and the frequency of accompanying myofascial pain syndrome in the breast cancer patients.

This study is designed as cross sectional- single centered and single blind. It is planned to include 110 breast cancer patients who had undergone the treatments as mastectomy, breast conserving surgery, lymph node dissection, sentinele lymph node biopsy or radiotherapy aged between 18-75 years-old, visiting our oncological rehabilitation outpatient clinic August 2023 through May 2024.

Patients will be divided into 2 groups according to the stage of lymphedema. It is known that pathophysiological changes develop even if there is no visible lymphedema in patients undergoing surgery and/or radiotherapy for breast cancer. There is a lifetime risk of developing lymphedema, so these patients are considered as Stage 0 (latent) . The patients with less than 3 cm difference between the circumference measurements of upper extremities will be included in the 1st group.( Stage 0) (n=55) Patients who have more than 3 cm difference between the circumference measurements of upper extremities and those with Stage 1,2 or 3 lymphedema will be included in the second group (n=55) The frequency of myofascial pain syndrome will be determined by the diagnostic criterias in both groups. The trigger points in trapezius, infraspinatus, serratus anterior, latissimus dorsi and pectoralis major muscles will be examined and the pain-pressure threshold values will be measured with an algometer.

For the evaluation of upper extremity function and quality of life following measurement tools will be utilized in both groups: Hand-grip test with a dynamometer, goniometric measurement of range of motion (ROM) of shoulder joint, VAS numerical scales, LYMQOL and DASH questionnaires.

Data analysis will be performed by using the Statistical Package for the Social Sciences (SPSS, version 20.0, IBM Corp., Armonk, NY, USA).

ELIGIBILITY:
Inclusion Criteria :

* Breast cancer patients aged between 18-75 who had undergone the treatments as mastectomy, breast conserving surgery, lymph node dissection, sentinele lymph node biopsy or radiotherapy providing a written consent to participate in the study

Exclusion Criteria :

* Patients who do not agree to participate the study
* Patients who had signs of active infection as lymphangitis, cellulitis, fungus
* Bilateral breast cancer patients
* Uncontrolled Psychiatric illness

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female Breast Cancer Patients
Study Population: Breast Cancer patients aged between 18-75 years old, who had undergone the treatments as mastectomy, breast conserving surgery, lymph node dissection, sentinele lymph node biopsy or radiotherapy visiting our oncological rehabilitation outpatient clinic between August 2023 and May 2024.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
The Evaluation of Trigger Points | 3 days
  Trigger points in trapezius, infraspinatus, latissimus dorsi, pectoralis major, serratus anterior muscles will be detected bilaterally by physical examination. Algometer (Wagner Force Dial FDK 20) will be used for pain pressure threshold measurement of detected trigger points. Then, the distribution of the trigger points, their frequency and threshold values according to the algometer will be compared between the individual affected-insured extremities and between the groups.
Clinical Diagnostic Criteria of Myofascial Pain Syndrome | 3 days
  Major criteria: 1. The patient's complaint of regional pain 2. Referred pain and sensory change in the specific area of the muscle by palpation of the trigger point 3. Presence of palpable taut band 4. Presence of palpable and tender points along the length of the taut band 5. Restriction of ROM in the area of the affected muscle Minor criteria: 1. Pain/sensory change with pressure palpation of the trigger point 2. Local twitch response with palpation/injection of the trigger point in the taut band 3. Reduction of pain by inactivation (injection or stretching of the muscle) of the trigger point 5 major and at least 1 minor criteria are required for clinical diagnosis

SECONDARY OUTCOMES:
Hand Grip Test | 3 days
  The purpose of this test is to test the maximum isometric contraction strength of the hand and forearm muscles. A hand grip dynamometer (Jamar) will be used for the test. While the patient is sitting in the chair, the elbows will be close to the body and at 90 degree flexion, the wrist will be in a neutral position. The patient will be asked to grasp the dynamometer and squeeze it as hard as she can, and the average of 3 measurements made with an interval of 5 minutes. The test will be repeated for both upper extremities separately.
Range of motion of shoulder joint | 3 days
  Goniometric measurements will be made for both upper extremities, and the average of 3 consecutive measurements will be taken.
VAS | 3 days
  Shoulder pain, feeling of tension and heaviness on the affected arm will be evaluated separately by numerical scale.
Quick-DASH (The Disabilities of the Arm, Shoulder and Hand) | 3 days
  The quick DASH questionnaire which has proven reliable and valid in breast cancer and lymphedema patients in Turkish population, will be used to evaluate the quality of life related to upper extremity function.
LYMQOL-arm (Lymphedema Quality of Life -arm) | 3 days
  Lymphedema Quality of Life Scale-Arm Turkish form will be used. The lymphedema-specific quality of life scale was developed specifically for the upper extremity and its reliability and validity were proven in Turkish population.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Bahar Özdemir, Principal Investigator
Locations (1):
- Sultan 2. Abdulhamid Han Training and Research Hospital, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Undecided